CLINICAL TRIAL: NCT04855305
Title: Optimizing and Standardizing 129Xe Gas Exchange MRI to Visualize Regional Therapy Response in Interstitial Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital Medical Center, Cincinnati (Other); University of Cincinnati (Other); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00107570; R01HL126771 (NIH)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Interstitial Lung Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with Interstitial Lung Disease (Active Comparator)
  Interventions: Drug: Hyperpolarized 129Xe
- Healthy Volunteers (Active Comparator)
  Interventions: Drug: Hyperpolarized 129Xe

INTERVENTIONS:
Drug: Hyperpolarized 129Xe — Hyperpolarized 129Xe will be administered in multiple doses in volumes that are tailored to the participant's total lung capacity (TLC) followed by a breath hold of up to 15 seconds.

SUMMARY:
The purpose of this multi-centered, NIH-sponsored study is to to develop an optimal protocol for using noninvasive 129Xe gas exchange MRI to detect changing disease activity in interstitial lung diseases (ILDs).

ELIGIBILITY:
Inclusion/Exclusion Criteria for Healthy Volunteers

Inclusion Criteria: Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Outpatients of either gender, age greater than or equal to 18 years
2. Willing and able to give informed consent and adhere to visit/protocol schedules (Consent must be given before any study procedures are performed.)
3. Subject has no diagnosed pulmonary conditions
4. Subject has not smoked in the previous 5 years
5. Smoking history, if any, is less than or equal to 5 pack-years
6. No history of using other inhaled products more than 1 time per week for > 1 year

Exclusion Criteria: Subjects presenting with any of the following will not be included in the trial:

1. Subject is less than 18 years old
2. MRI is contraindicated based on responses to MRI screening questionnaire
3. Subject is pregnant or lactating
4. Resting oxygen saturation on room air <90%
5. Respiratory illness of a bacterial or viral etiology within 30 days of MRI
6. Subject has history of any known ventricular cardiac arrhythmia
7. Subject has history of cardiac arrest within the last year
8. Subject does not fit into Xe vest coil used for MRI 129
9. Subject cannot hold his/her breath for 15 seconds
10. Subject deemed unlikely to be able to comply with instructions during imaging
11. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Inclusion/Exclusion Criteria for Subjects with Interstitial Lung Disease

Inclusion Criteria: Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the trial:

1. Outpatients of either gender, age greater than or equal to 18 years
2. Willing and able to give informed consent and adhere to visit/protocol schedules (Consent must be given before any study procedures are performed.)
3. Clinical diagnosis of Interstitial Lung Disease made by a board certified pulmonologist using established criteria. We will not exclude individuals based on ILD type or severity of disease with the exception of the below criteria

Exclusion Criteria: Subjects presenting with any of the following will not be included in the trial:

1. Subject is less than 18 years old
2. MRI is contraindicated based on responses to MRI screening questionnaire
3. Subject is pregnant or lactating
4. Resting oxygen saturation <90% on supplemental oxygen
5. Respiratory illness of a bacterial or viral etiology within 30 days of MRI
6. Subject has history of any known ventricular cardiac arrhythmia.
7. Subject has history of cardiac arrest within the last year
8. Subject does not fit into Xe vest coil used for MRI 129
9. Subject cannot hold his/her breath for 15 seconds
10. Subject deemed unlikely to be able to comply with instructions during imaging
11. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Thoracic cavity volume measured in liters. | 4 years
RBC/barrier signal ratio (unitless). | 4 years
Coefficient of repeatability of RBC/barrier signal ratio (unitless). | 4 years
Echo time to separate RBC and barrier signals by 90 degrees (ms). | 4 years
Population-wide RBC/barrier signal ratio (unitless). | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mammarappallil, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
A major focus of this work is sharing and dissemination of the image acquisition and analysis methods we develop as well as standard operating procedures for 129Xe MRI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: A major focus of this work is sharing and dissemination of the image acquisition and analysis methods we develop as well as standard operating procedures for 129Xe MRI. In all instances we will adhere to the NIH Sharing Policies and Related Guidance on NIH-Funded Research Resources for Recipients of NIH Grants and Contracts on Obtaining (https://grants.nih.gov/policy/sharing.htm) and Disseminating Biomedical Research Re-sources (issued December 1999). However, we intend to greatly exceed these requirements, making as much of our work freely available to the broader research community either before, or immediately after publication of manuscripts, as well as through PubMedCentral. While we we will provide relevant protocols upon request at any time, we further intend to pursue several proactive data sharing mechanisms.
Access Criteria: We are committed to making de-identified datasets and image analysis available to to qualified investigators. When required scientifically, data including identifiers will be shared under an agreement that provides for: (1) a commitment to using data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data appropriately; and (3) a commitment to destroying or returning the data after analyses are completed.